CLINICAL TRIAL: NCT05146843
Title: The Impact of Chronic Mitochondrial Antioxidant (MitoQ) Supplementation on Cardiovascular Toxicity Induced by Doxorubicin-Based Adjuvant Chemotherapy in Breast Cancer Patients: Randomized Clinical Trial
Brief Title: The Impact of Chronic Mitochondrial Antioxidant Supplementation on CardiovascularToxicity in Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: InCor Heart Institute (Other); Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Allan Robson Kluser Sales, PhD, D'Or Institute for Research and Education
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 48347821.8.0000.5249
Record Dates: First submitted 2021-11-24; First posted 2021-12-07 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Breast Neoplasms
Keywords: Breast Cancer; Doxorrubicin; Mitoquinone; Cardiotoxicity; Peripheral vascular function
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity | interventions — mitoquinone

STUDY DESIGN:
Intervention Model Description: Clinical, randomized, double-blind, placebo-controlled trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mitoquinone (Experimental): MitoQ, 20 mg per day for three months
  Interventions: Drug: Mitoquinone
- Placebo (Placebo Comparator): Placebo, 20 mg per day for three months
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mitoquinone — Mitoquinone pill, 20 mg/day
  Other Names: MitoQ
  Arms: Mitoquinone
Other: Placebo — Placebo pill, 20 mg/day
  Arms: Placebo

SUMMARY:
Investigate the protective effect of chronic MitoQ supplementation on cardiovascular toxicity induced by doxorubicin-based adjuvant chemotherapy in breast cancer patients.

DETAILED DESCRIPTION:
Test the hypothesis that chronic MitoQ supplementation in breast cancer patients treated with doxorubicin prevents:

1. increased mitochondrial oxidative stress;
2. the increase in cardiac markers (B-type natriuretic peptide and troponin I);
3. changes in left ventricular deformity (speckle tracking, strain) and reduction in LVEF;
4. endothelium-dependent dysfunction of peripheral vascular beds;
5. the increase in endothelial microvesicles;
6. the increase in material stiffness;
7. the elevation of central blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old, diagnosed with breast cancer (ductal, lobular and mixed carcinoma), in stage 1-3, with indication for the adjuvant AC-T therapeutic scheme, doxorubicin (60 mg/m2) plus cyclophosphamide, will be considered eligible for the study (600 mg/m2) in the regimen of 1 cycle every 21 days, followed by weekly taxane for 12 cycles.

Exclusion Criteria:

* Patients with metastasis, severe lymphedema, renal failure, acute myocardial infarction, heart failure, stroke and chronic liver disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-06-02 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-12-02 (Estimated)

PRIMARY OUTCOMES:
Changes of the left ventricular deformity and reduction in left ventricular ejection fraction | 3 Months
  Cardiac function changes (Strain and Simpson's monoplanar)

SECONDARY OUTCOMES:
Systemic markers of oxidative stress | 3 Months
  Mitochondrial oxidative stress; Cardiac markers (B-type natriuretic peptide and troponin I);
Endothelium-dependent dysfunction of peripheral vascular beds | 3 Months
  changes in the endothelium-dependent function of peripheral vascular beds
Arterial stiffness | 3 Months
  Increase in the arterial stiffness
Central blood pressure | 3 Months
  Alterations on the central blood pressure
Physical capacity | 3 Months
  Reduction in the peak oxygen uptake

CONTACTS AND LOCATIONS:
Overall Officials: Allan Kluser Sales, PhD, Principal Investigator — D'Or Institute of Research and Education